CLINICAL TRIAL: NCT00779935
Title: Baseline Serum Vascular Endothelial Growth Factor (VEGF) Concentration as Predictive Factor of Response to Infliximab (Remicade) Therapy in Patients With Active Ankylosing Spondylitis Despite Conventional Treatment: a Multicenter Pilot Study
Brief Title: Growth Factor Concentration to Predict an Ankylosing Spondylitis Patient's Response to Infliximab (Study P04041)(COMPLETED)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P04041
Record Dates: First submitted 2008-10-23; First posted 2008-10-24 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Spondylitis, Ankylosing
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Remicade (Experimental): Remicade will be given at Weeks 0, 2, and 6 and then every 8 weeks up to Week 54.
  Interventions: Biological: Remicade

INTERVENTIONS:
Biological: Remicade — Remicade will be given at Weeks 0, 2, and 6 and then every 8 weeks up to Week 54.
  Other Names: Infliximab; SCH 215596

SUMMARY:
This is a Phase 4, multi-center, open-label, one-arm, pilot study in patients with active ankylosing spondylitis refractory to conventional treatment. Remicade will be given at Weeks 0, 2, and 6 and then every 8 weeks up to Week 54. The number of patients showing ASAS-20 clinical response at Week 14 will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ankylosing spondylitis proven by appropriate diagnostic methods (according to New York criteria).
* Refractory disease defined by failure of at least 2 non-steroidal anti-inflammatory drugs (NSAIDs) during a 3-month period and failure of sulfasalazine in subjects with associated peripheral arthritis.
* Active disease defined by:

  * sustained BASDAI of at least 40 on a 0-100 scale and
  * expert opinion based on clinical features.
* Age between 18 and 70 years.
* Subjects using NSAIDs and/or sulfasalazine must have been on a stable dose for at least 4 weeks prior to study initiation, and may continue medication during the treatment period, but the dose must not be increased above the baseline.
* Subjects must be capable to demonstrate their willingness to participate in the study and comply with its procedures by signing a written informed consent.
* Men and women of childbearing potential (includes women who are less than 1 year postmenopausal and women who become sexually active) must be using an acceptable method of birth control (eg, hormonal contraceptive, medically prescribed IUD, condom in combination with spermicide) or be surgically sterilized (eg, hysterectomy or tubal ligation).
* Subjects must understand and be able to adhere to the dosing and visit schedules.

Exclusion Criteria:

* Subject with moderate or severe heart failure (NYHA class III/IV).
* Remicade must not be given to subjects with a history of hypersensitivity to infliximab, to other murine proteins, or to any of the excipients.
* Subjects with pre-existing or recent onset of central nervous system demyelinating disorders.
* Age <18 or >70 years.
* Pregnant women, nursing mothers.
* Subjects who are incapacitated, largely or wholly bedridden or confined to a wheelchair, and who have little or no ability for self-care.
* Subjects who have any current systemic inflammatory condition with signs and symptoms that might confound the evaluations of benefit from infliximab therapy.
* Prior administration of infliximab or any other therapeutic agent targeted at reducing TNF (eg, Etanercept, pentoxifylline, thalidomide or anti-CD4+ antibody).
* Current treatment with systemic corticosteroid.
* Treatment with any investigational drug within the previous 3 months.
* History of known allergies to murine proteins.
* Subjects having active or inactive tuberculosis (TB). All subjects must be evaluated for both active and inactive ('latent') TB. This evaluation should include a detailed medical history with personal history of TB or possible previous contact with TB and previous and/or current immunosuppressive therapy. Appropriate screening tests (ie, tuberculin skin test and chest x-ray) should be performed in all subjects.
* Serious infection, such as sepsis, abscesses, hepatitis, pneumonia, pyelonephritis in the previous 3 months. Less serious infections in the previous 3 months, such as acute respiratory tract infection (colds) or uncomplicated urinary tract infection need not be considered exclusions at the discretion of the treating physician.
* History of opportunistic infections such as herpes zoster within 2 months of study initiation. Evidence of active CMV, active pneumocystis carinii, drug resistant atypical mycobacterium, etc.
* Documented HIV infection.
* Current signs or symptoms of severe, progressive or uncontrolled renal, hepatic, hematologic, endocrine, pulmonary, cardiac, neurological, or cerebral disease.
* Any currently known malignancy or pre-malignant lesions or any history of malignancy within the past 5 years (except non-melanoma skin cancer and surgically cured cervical cancer).
* Subjects with alcoholism, alcoholic liver disease, or other chronic liver disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2004-10-01 (Actual); Primary Completion 2005-10-01 (Actual); Study Completion 2007-02-01 (Actual)

PRIMARY OUTCOMES:
To investigate whether baseline serum VEGF concentration predicts ASAS-20 clinical response to infliximab at Week 14. | Week 14

SECONDARY OUTCOMES:
To detect clinical response rates at Weeks 2, 6, 14, 30, 54, and at Follow-up Visit 2, which is 6 months after completion of study treatment. | Weeks 2, 6, 14, 30, 54 and 6 months afterwards
To measure the duration of response | Weeks 2, 6, 14, 30, 54 and 6 months afterwards
To detect the percent of patients reaching partial response | Weeks 2, 6, 14, 30, 54 and 6 months afterwards
To measure the duration of partial response | Weeks 2, 6, 14, 30, 54 and 6 months afterwards

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html